CLINICAL TRIAL: NCT00236041
Title: A Double-Blind, Placebo-Comparison Study to Evaluate the Efficacy and Safety of ACTIQ® (Oral Transmucosal Fentanyl Citrate [OTFC®]) Treatment for Opioid-Tolerant Children and Adolescents With Breakthrough Pain
Brief Title: Efficacy/Safety Study of ACTIQ® for Opioid-Tolerant Children and Adolescents With Breakthrough Pain (BTP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: C8278b/202/BP/US-CA
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Cancer; Breakthrough Pain
Keywords: Breakthrough Pain; Cancer; Sickle Cell; Severe Burns; Children; Adolescents; Analgesia; Sickle Cell Disease; Non-Cancer
MeSH Terms: conditions — Neoplasms; Breakthrough Pain; Burns; Agnosia; Anemia, Sickle Cell | interventions — Fentanyl

INTERVENTIONS:
Drug: ACTIQ®

SUMMARY:
The primary objective of the study is to evaluate the efficacy of ACTIQ treatment for the management of breakthrough pain (BTP) compared to placebo treatment in children with cancer and non-cancer pain who are receiving around-the-clock (ATC) opioid therapy and who require additional therapy for BTP episodes. This will be determined by the analysis of the pain intensity (PI), measured by the Faces Pain Scale-Revised (FPS-R) administered 15 minutes after the start of each unit of study drug with an optimal ACTIQ dosage.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy of ACTIQ treatment for the management of breakthrough pain (BTP) compared to placebo treatment in children with pain who are receiving around-the-clock (ATC) opioid therapy and who require additional therapy for BTP episodes. This will be determined by the analysis of the pain intensity (PI), measured by the Faces Pain Scale-Revised (FPS-R) administered 15 minutes after the start of each unit of study drug with an optimal ACTIQ dosage.

The secondary objectives are:

* to evaluate the characteristics of BTP in children with pain, including their response to treatment
* to evaluate the efficacy of ACTIQ treatment compared to placebo treatment for these children with regard to time to adequate analgesia by utilizing a stop watch to measure the time for each unit of study drug in the double blind phase
* to evaluate the efficacy of ACTIQ treatment compared to placebo treatment for these children by assessing the occurrence of inadequate analgesia as assessed by the use of rescue medication
* to evaluate the efficacy of ACTIQ treatment compared to placebo treatment for these children by assessing the numbers of patients who withdraw from the study because of inadequate analgesia
* to evaluate the efficacy of ACTIQ treatment compared to placebo treatment for these children by assessing the duration of analgesic effect by using the FPS-R administered at approximately 30, 45, and 60 minutes after the start of each unit of study drug after an optimal dosage is obtained
* to determine the distribution of optimal doses of ACTIQ treatment for these children by age group (3 to under 6 years, 6 to under 11 years, and 11 to under 16 years)
* to establish a safe and effective titration scheme for ACTIQ in these children during the open label phase
* to evaluate the safety of ACTIQ treatment for these children through the assessment of adverse events, clinical laboratory assessments (serum chemistry and hematology), vital sign measurements (including blood pressure, heart rate, and respiration rate), hemoglobin-oxygen saturation level (SpO2, measured via pulse oximetry), electrocardiograms (ECGs), physical examinations, and level of sedation (measured by the University of Michigan Sedation Scale [UMSS])
* to characterize the pharmacokinetics profile of ACTIQ (fentanyl citrate) in these children
* to investigate the exposure and efficacy relationship between plasma concentration of fentanyl and clinical measures of analgesia

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of the parent or legal guardian and patient assent, when appropriate, is obtained. (Lack of assent cannot be overturned.)
2. The child is aged 3 to under 16 years and weighs at least 15 kg.
3. The child must be using ATC opioid therapy for pain associated with cancer and be opioid-tolerant. NOTE: This requirement is defined as the patient receiving at least 1 mg/kg/day or 40 mg/day or more of oral morphine (or an equi-analgesic dosage of another opioid) or at least 25 mcg/hour of transdermal fentanyl for at least 7 days, (ATC opioid therapy may be administered as patient-controlled analgesia [PCA]).
4. The child must be experiencing episodes of BTP (defined as a transient flare of pain that requires a bolus of medication as treatment) as follows:

   1. patients with cancer must be experiencing an average of at least 1 BTP episode a day.
   2. patients with non-cancer related pain must be experiencing an average of 2 BTP episodes a day.
5. The child has an average daily pain score of 6 or less (of 10) on the FPS-R.
6. Girls who are postmenarche or sexually active must have a negative urine pregnancy test prior to the baseline visit, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implanted, or injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence.
7. The child, in the opinion of the investigator, is able to administer ACTIQ treatment effectively (ie, adequately moving the unit around in the mouth and sucking, not biting, the unit).
8. The child must be an inpatient.

Exclusion Criteria:

1. The child has pain uncontrolled by therapy, as determined by the investigator, that could adversely impact the safety of the patient or could be compromised by treatment with ACTIQ.
2. The child has known or suspected hypersensitivities/allergies or other contraindications to any ACTIQ component.
3. The child has received monoamine oxidase inhibitors (MAOIs) within 14 days before the first ACTIQ treatment.
4. The child has moderate to severe oral mucositis.
5. The child has a neuromuscular disease, significant renal impairment, or significant hepatic impairment as determined by the investigator.
6. The child has any other medical condition or is receiving concomitant medication/therapy that would, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise data collection.
7. The child has received any experimental drug/therapy within 14 days of the first ACTIQ treatment. NOTE: Children may not be participating concurrently in another study when the other study requires experimental drug therapy.
8. A child's exacerbations of pain are only associated with medical procedures (such as radiation therapy, wound dressing, and bone marrow aspiration).
9. The child is receiving any other treatment that, in the opinion of the investigator, could interfere with the pain response.
10. For a female patient of childbearing potential: is pregnant or lactating. (Any female patient becoming pregnant during the study will be withdrawn from the study.)
11. The child has, in the opinion of the investigator, developmental delay that would interfere with the use of ACTIQ therapy.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38
Dates: Start 2004-04; Study Completion 2006-08

PRIMARY OUTCOMES:
Pain intensity differences as measured by the FPS-R

SECONDARY OUTCOMES:
Time to adequate analgesia
Duration of analgesia
Percentage of BTP episodes requiring rescue medication, or for which oversedation occurs
Amount of rescue medication
Distribution of optimal doses

CONTACTS AND LOCATIONS:
Overall Officials: John Messina, Pharm D, Study Director — Cephalon, Inc.
Locations (31):
- United States (30):
  - Children's Hospital of Arkansas, Little Rock, Arkansas
  - UCLA Pediatric Pain Program, Los Angeles, California
  - Childrens Hospital of Orange, Orange, California
  - Lucille Packard Childrens Hospital, Palo Alto, California
  - Connecticut Childrens Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Childrens Clinic, Jacksonville, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Scottish Rite Children's Medical Center, Atlanta, Georgia
  - Kapi'olani Medical Center, Honolulu, Hawaii
  - Children's Memorial Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - University Hospitals of Iowa, Iowa City, Iowa
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - SUNY Upstate Medical University, Syracuse, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Milton S Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Vanderbilt University Medical, Nashville, Tennessee
  - Children's Cancer and Blood Disorders Center, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- San Jorge Childrens Medical, San Juan, Puerto Rico